CLINICAL TRIAL: NCT03550261
Title: Salt Wasting, Hydro-sodium Balance and Fludrocortisone Requirement in Congenital Adrenal Hyperplasia
Acronym: NaCAH
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI17028J
Record Dates: First submitted 2018-04-05; First posted 2018-06-08 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Congenital Adrenal Hyperplasia (CAH)
Keywords: CAH; Salt-wasting; LC-MSMS; plasma and urine steroid profile; Fludrocortisone
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — For blood samples, the biochemistry laboratory of each investigating centre will centrifuge all blood samples, collect the plasma and transfer it into a new tube on which the corresponding labels will be affixed.
  The tubes will be frozen at -20° C in a freezer at a specific location where the tubes with the same identification number (blood and urine sample from the same child) will be grouped.
  The urinary samples (H0, H48, M1, M3 and M6) collected on a gauze compress will arrive at the laboratory of each centre in tubes already labelled (sterile urine jar) and will be frozen directly at -20° C with the tubes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Congenital adrenal hyperplasia (CAH) in its classic neonatal form with severe salt-wasting represents a challenge for pediatric endocrinologists in order to maintain sodium balance, especially as the physiopathology and optimal therapeutic management of this urinary salt loss remain poorly studied, particularly during the neonatal period.

The human kidney presents the characteristic of being immature at birth with a functional tubulopathy associating sodium wasting and difficulty to concentrate urine, in connection with a transient renal resistance to aldosterone action, which is exacerbated in case of CAH by insufficiency of aldosterone production.

The objective of project is therefore to study the secretion profiles of plasma and urinary steroids in neonates with classical salt-wasting form of CAH before treatment and under treatment with Fludrocortisone and Hydrocortisone during the first months of life, using an advanced technology: LC-MSMS (Liquid chromatography coupled with tandem mass spectrometry). The study of the existence of a correlation between plasma and urinary steroid profiles will also make it possible to subsequently consider simplified medical follow-up for these patients.

This project will lead to a better understanding of sodium handling and steroid secretion and excretion profiles in CAH neonates, in order to improve the therapeutic management of mineralocorticoid replacement in these patients.

DETAILED DESCRIPTION:
Congenital adrenal hyperplasia in its severe salt-wasting form is a challenge in order to maintain sodium balance. The pathophysiology of this impaired sodium balance is still poorly investigated as well as its therapeutic management, notably in the neonatal period. Consensus practice guidelines have been established for hydrocortisone replacement therapy, in order to maintain negative feedback on the pituitary-adrenal axis to prevent from virilization and excessive growth velocity. However, mineralocorticoid substitution and sodium supplementation is currently empirically adapted based on weight gain and renin levels. There is significant need for improvement of this essential part of CAH treatment. Particularly, CAH patients have higher risk of adverse cardio-vascular outcomes, which could relate to an excessive glucocorticoid and/or mineralocorticoid exposure in early infancy rather than to the genotype of the patient.

A clinical human study in classical CAH neonates, using Liquid Chromatography coupled to tandem Mass Spectrometry LC-MS/MS technology will assess prospectively plasma and urinary steroid profiling (precursors and substitute hormones, notably Fludrocortisone dosages) during the first six months of life, before and under treatment; and in correlation with genotype.

Thirty neonates (boys and girls) diagnosed with a severe form of CAH and followed in one of the 5 following French reference tertiary centers: Robert Debré Hospital, Paris; Necker Hospital, Paris; Bicetre Hospital, Le Kremlin-Bicetre; Trousseau Hospital, Paris; Lyon Hospital, , will be included in the study and will be followed for a period of six months. The duration of inclusion will be 24 months.

Genotyping will be processed for all children in Lyon.This project will lead to a better understanding of sodium handling and steroid secretion and excretion profiles in CAH neonates, in order to improve management of mineralocorticoid replacement.

ELIGIBILITY:
Inclusion Criteria:

* Newborns with confirmation or strong suspicion of diagnosis of congenital adrenal hyperplasia:
* Newborns with abnormal differentiation of the external genitalia, without palpable gonad at birth and high 17 OHP plasma level
* Newborns diagnosed with antenatal CAH,
* Newborns diagnosed at birth with CAH (due to parents at risk of transmission of the disease),
* Newborns diagnosed by systematic screening for 17 OHP on the 3rd day of life (thus having a high dosage of 17 OHP), confirmed by a second sample.

For all these patients the diagnosis of CAH will have to be confirmed secondarily by molecular biology.

Exclusion Criteria:

* Newborn with an anomaly of sexual differentiation from another origin,
* Newborn already under treatment with Fludrocortisone and/or Hydrocortisone.

Ages: 1 Day to 15 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborns (boys and girls) diagnosed with a neonatal form of CAH and followed up in one of the following 5 French reference centres: Robert Debré Hospital, Paris; Necker Hospital, Paris; Bicêtre Hospital, Le Kremlin-Bicêtre; Trousseau Hospital, Paris; Femme-Mère-Enfant Hospital, Lyon.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
Plasma LC-MSMS dosages | 48 hours
  Determine if a correlation exist between plasma and urinary steroid profile by LC-MSMS and genotype before treatment, and if there exist a correlation to the Fludrocortisone dose after 48h of treatment
Urinary LC-MSMS dosages | 48 hours
  Determine if a correlation exist between plasma and urinary steroid profile by LC-MSMS and genotype before treatment, and if there exist a correlation to the Fludrocortisone dose after 48h of treatment

SECONDARY OUTCOMES:
Plasma LC-MSMS dosages | day1, day2, 1 month, 3 months and 6 months
  Steroid profiles will be compared between urine and plasma to search for a correlation
Urinary LC-MSMS dosages | day1, day2, 1 month, 3 months and 6 months
  Steroid profiles will be compared between urine and plasma to search for a correlation

CONTACTS AND LOCATIONS:
Overall Officials: Martinerie Naetitia, PHD, Principal Investigator — APHP
Locations (1):
- Hôpital Robert Debré, Paris, France